CLINICAL TRIAL: NCT04278014
Title: Evaluation of Ultrasound Guided Continuous Sciatic Block Nerve With a Longitudinal Approach in the Management of Vascular Pain in Critical Ischemia of Lower Limbs Patients : Prospective Descriptive Study of Exploratory Cohort
Brief Title: Continuous Sciatic Block Nerve in the Management of Vascular Pain in Critical Ischemia of Lower Limbs Patients
Status: Completed | Type: Observational
Sponsor: Universidad de Antioquia (Other)
Responsible Party: Sponsor
Other Study IDs: UdeA1006
Record Dates: First submitted 2020-02-18; First posted 2020-02-20 (Actual); Last update posted 2021-05-05 (Actual); Status verified 2021-02

CONDITIONS: Critical Limb Ischemia
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: ultrasound-guided continuous sciatic block with longitudinal approach — ultrasound-guided continuous sciatic block with longitudinal approach

SUMMARY:
Critical limb ischemia (CLI) is associated with severe pain that is a therapeutic challenge whit therapeutic limits for the use of conventional analgesics medications. ultrasound-guided continuous sciatic block (CCBN) is strategy effective and safe to consider in this patients.

This prospective descriptive exploratory cohort study evaluates CCBN as a effective therapeutic tools for patients whit (CLI)

DETAILED DESCRIPTION:
Critical limb ischemia is the final stage of peripheral vascular disease identified by resting pain greater than 2 weeks with ulcers or gangrene in 1 or both extremities. Pain relief is a therapeutic challenge due to its severity, which significantly affects the quality of life, and the comorbidities that occur frequently in these patients, which limits the use of analgesics medications. Regional techniques can play an important role as they are safe and effective in analgesic management . Within these we find the ultrasound guided continuous sciatic block as a strategy to consider in the periods of exacerbation of pain, as a bridge to a palliative or resolutive management.

Prospective descriptive exploratory cohort study.

Patients with a diagnosis of critical ischemia of the lower limb with severe pain and side effects of opioids will be included. A continuous ultrasound-guided sciatic nerve block with longitudinal approach will be performed, with no anti-aggregation or anticoagulation suspension, continuing with an infusion of Bupivacaine 0.1%

The primary outcome will be numerical pain rating scale (NPrs) and secondary outcome Pinprick test, catheter duration, opioid consumption reduction and side effects to it.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of critical ischemia of the lower limb with severe pain and side effects of opioids

Exclusion Criteria:

* Under 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of critical ischemia of the lower limb with severe pain and side effects of opioids over 18 years old who accept the interventional technique
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Pain level measurement with Numeric Rate Score (NRS) | 5 days
  0-10 where 0 means no pain and 10 means maximum possible pain

SECONDARY OUTCOMES:
Pinprick test | 5 days
  evaluation of superficial sensitivity in S1 dermatome positive or negative
catheter duration | 5 days
  number of days in which the catheter is functional
opioid consumption reduction | 5 days
  opioid consumption in morphine equivalence
Delirium | 5 days
  minimental test score from 0 to 30 points. Delirium positive for less than 24
Nauseas and Vomit | 5 days
  yes or not present

CONTACTS AND LOCATIONS:
Locations (2):
- Colombia (2):
  - hospital universitario San Vicente Fundacion, Medellín, Antioquia
  - Adriana Cadavid, MD, Medellín, Antiquia

IPD SHARING:
Plan to Share IPD: No